CLINICAL TRIAL: NCT02907411
Title: Quadrivas Therapy® to Reduce Lipedema Subcutaneous Adipose Tissue (QUADRIVAS)
Acronym: QUADRIVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Hanger Clinic: Prosthetics & Orthotics (Other); Quadrivas Therapy Clinic & Academy Amsterdam (Unknown)
Responsible Party: Principal Investigator, KHerbst, Associate Professor, TREAT Program Director, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1607696709
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Lipedema
Keywords: Quadrivas; Veins; Lipedema; Lymphedema
MeSH Terms: conditions — Lipedema; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quadrivas Therapy (Experimental): Hands on therapy to improve all aspects of fat tissue including the vessels within. Each of 7 subjects receive 12 treatments in one month time.
  Interventions: Other: Quadrivas Therapy

INTERVENTIONS:
Other: Quadrivas Therapy — Quadrivas therapy will be applied to subjects. Quadrivas therapy is a intensive massage therapy for different tissues. Subjects will receive 12 treatments. The first lasting 2.5 hours and the remaining 11 lasting 1.5 hours.

SUMMARY:
Quad Rivas Therapy has been developed by Alyna Eekma from the Netherlands for over thirteen years; anecdotally she has been able to significantly reduce lipedema SAT in women with Stage 1 and 2 lipedema, and can reduce lipedema SAT by 80% in women with Stage 3 lipedema. The study will last for one month, for a total of 12 treatments per subject, seven subjects total, to see if there is a change in percent body fat percentage over the course of these treatments.

DETAILED DESCRIPTION:
Lipedema

According to an epidemiological study by Földi E and Földi M, lipedema affects 11% of the female population. Rarely, men with hypogonadism, growth hormone deficiency, or liver disease may develop lipedema. Drs. Allen and Hines from the Mayo clinic defined lipedema in 1940 and shortly thereafter provided the diagnostic criteria for lipedema:

1. Almost exclusive occurrence in women developing by the third decade of life
2. Bilateral and symmetrical nature with minimal involvement of the feet, resulting in an ''inverse shouldering'', ''bracelet'' or "cuff" effect at the ankle
3. Minimal pitting edema (non-pitting edema is present)
4. Pain, tenderness, and easy bruising
5. Persistent enlargement despite elevation of the extremities or weight loss.
6. Increased vascular fragility; easy bruising

There are three stages of lipedema Stage 1: Normal skin surface with enlarged hypodermis Stage 2: Uneven skin with a peau d'orange or mattress-like texture with larger mounds of tissue the size of a walnut or apple including the formation of lipomas and angiolipomas, and larger indentations in the fat Stage 3: Much larger mounds or huge lobules of tissue occurs causing deformations especially around the knees

Progression to lymphedema, called lipolymphedema (Stage 4) can develop during any Stage but most commonly occurs in people with Stage 3. Obesity can occur along with lipedema especially in Stage 3. Lifestyle improvements should always be considered for obesity associated with lipedema but lifestyle is not the cause of lipedema nor the cure.

Women with lipedema have an obvious disparity between the larger quantity of gynoid distributed painful fat on the lower body (hips, buttocks, legs) compared to the trunk, head and face resulting in a low waist to hip ratio (WHR). The disparity results from the failure of lipedema SAT to reduce in response to extreme caloric restriction, including bariatric procedures, or intensive daily exercise. It is unclear why there is a drive to maintain lipedema SAT on the body. The SAT begins in typical gynoid locations (hips, buttocks, legs) and few women with lipedema have diabetes or metabolic syndrome suggesting that the lipedema SAT may be protective against cardiovascular disease similar to gynoid fat. However, in addition to being cosmetically devastating to many women, lipedema fat increases the risk of development of mobility issues, joint damage, chronic pain and lymphedema.

Quad Rivas Therapy®

The Quad Rivas Therapy® is a deep tissue "hands on" touch therapy of SAT which treats the body as an anatomical and physiological unit - all areas containing SAT are treated with a focus to improve functioning of blood vasculature, lymph vasculature, nerves, and the biomechanical system (muscle, tendons and fascia). The Quad Rivas Therapy® ensures these four systems are improved, but focuses on the vascular system. Tissues with decreased blood supply due to enlarged SAT mass, fibrosis or fascia disease need manipulation to be able to function properly again, allowing easy flow through the tissue. The Quad Rivas Therapy, therapist uses specialized grip techniques which enable the therapist to 'open' and 'unravel' tissues for an optimal blood supply. Another tissue technique, called the "hook technique" allows the therapist to ensure stimulation of blood flow. Blood vessels gain elasticity back, fibrosis in the veins resolves and the body is able to repair itself.

The Quad Rivas Therapy® theory is that during puberty under the influence of hormones, the lipedema SAT outgrows the ability of muscles to use and break down fat resulting in excess SAT mass. This in combination with vascular, especially venous, insufficiency, which affects many women at a young age, creates a progressive disease that generates a blockage in metabolism associated due to setting up a hypoxic environment for the fat cells. Stimulating the affected area with Quad Rivas Therapy®, focusing on getting vessels back in top condition ensures the disappearance of lipedema SAT.

Quad Rivas Therapy® results in the following:

1. Recovery of the walls of the veins;
2. Increased basal metabolic rate in muscles;
3. Improved condition of the connective tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory females of any race able to understand the consent process.
2. 19-70 years of age.
3. Diagnosis of lipedema Stage 1 or Stage 2 although early Stage 3 will be considered.
4. Weight stable for past three months per personal report of the subject.
5. Must be able to attend all 12 treatments and pre and post procedures

Exclusion Criteria:

1. Use of medications that might cause weight gain and prevent fat loss (e.g., second generation anti-psychotics, corticosteroids).
2. Current use of weight loss medications.
3. Tobacco or marijuana use which may alter inflammation in the body.
4. Pregnancy due to the risks associated with deep tissue treatment.
5. Two or more alcoholic beverages per day, chronically.

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09-01; Primary Completion 2017-03-18 (Actual); Study Completion 2017-03-18 (Actual)

PRIMARY OUTCOMES:
Full Body Fat Percentage | Baseline and 4 weeks
  Change in full body fat percentage after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Herbst, MD, PhD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - The Herbst Clinic, Tucson, Arizona
  - Clinical and Translational Sciences Research Center (CATS) at the University of Arizona, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared with investigators who submit a request